CLINICAL TRIAL: NCT06746857
Title: iTBS-Neurosplasticity for Female Youth With Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Fidel Vila-Rodriguez, MD, PhD, FRCPC, DFAPA, Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H22-02593
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accelerated iTBS (Experimental)
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — Bilateral dorsolateral prefrontal cortex Intermitten Theta Burst Stimulation to

SUMMARY:
TBC

DETAILED DESCRIPTION:
TBs

ELIGIBILITY:
Inclusion Criteria:

1. are assigned female sex at birth;
2. are 16yo to 24yo;
3. outpatients;
4. are competent to assent (those age 16-18) or consent to participate (those age 19-24);
5. have a Diagnostic and Statistical Manual of Mental Disorders Fifth edition (DSM 5) diagnosis of Major Depressive Episode by Mini-International Neuropsychiatric Interview (MINI) version 7.0.0 for participants aged 18-24 and Adolescents (MINI-KID) for participants aged 16-17;
6. have a score ≥ 18 on the Hamilton Depression Rating Scale (HDRS-17 item) or Depressive symptom severity as shown by a total Children's Depression Rating Scale Revised (CDRS-R) score 40;
7. have not changed dose or initiated a new regular antidepressant or antidepressant augmentation treatment(s) for 4 weeks prior to starting TMS treatment;
8. are able to adhere to the treatment schedule;
9. pass both the TMS and MRI adult safety screening questionnaires.

Exclusion Criteria:

1. have Moderate or Severe Substance Use Disorder (except tobacco) within the last three (3) months;
2. have a concomitant major unstable medical illness;
3. have active suicidal intent;
4. have not responded to 2 or more adequate trials of antidepressant medication in the current episode as meassured by the ATHF form
5. are pregnant or planning to become pregnant during the study period;
6. have a lifetime (MINI) diagnosis of any psychotic disorder;
7. have a MINI anxiety disorder or personality disorder assessed by a study investigator to be primary and causing greater impairment than MDE;
8. have previously had ECT or rTMS;
9. have any significant neurological disorder or any significant head trauma with clear radiological evidence of cerebrovascular injury on imaging.
10. have any intracranial implant (e.g., aneurysm clips) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed;
11. have history of epilepsy
12. are participating in standardized regular psychotherapy provided by a psychiatrist or a registered psychologist for less than 3 months prior to study entry or planning to start during the course of rTMS treatments;
13. have a clinically significant laboratory abnormality, in the opinion of the one of the principal investigators;
14. have a non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview);

Ages: 16 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale Depression | Four weeks
  Minimum score: 0; Maximum score: 52; higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Fidel Vila-Rodriguez, MD, PhD, FRCPC, DFAPA, Principal Investigator — University of British Columbia